CLINICAL TRIAL: NCT00079248
Title: UK Trial Of Hormone Replacement Therapy (HRT) In Women With A History Of Early Stage Breast Cancer
Brief Title: Hormone Replacement Therapy in Relieving Menopausal Symptoms in Postmenopausal Women With Previous Stage I or Stage II Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000355122; CRUK-HRT; EU-20112; ISRCTN29941643
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2005-06

CONDITIONS: Breast Cancer; Hot Flashes; Menopausal Symptoms; Osteoporosis
Keywords: osteoporosis; stage I breast cancer; stage II breast cancer; menopausal symptoms; hot flashes
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes; Osteoporosis | interventions — Progesterone; Estrogens, Conjugated (USP)

INTERVENTIONS:
Biological: therapeutic progesterone
Drug: conjugated estrogens

SUMMARY:
RATIONALE: Hormone replacement therapy may be effective in relieving symptoms of menopause, such as hot flashes, night sweats, and vaginal dryness, without causing a recurrence of breast cancer.

PURPOSE: This randomized clinical trial is studying hormone replacement therapy to see how well it works in relieving symptoms of menopause in postmenopausal women with previous stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare disease-free survival and overall survival of postmenopausal women with prior stage I or II breast cancer treated with hormone replacement therapy (HRT) vs nonhormonal alternatives to HRT.
* Compare relief of menopausal symptoms and quality of life of patients treated with these regimens.
* Compare cardiovascular and osteoporotic events in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, age (< 40 years vs ≥ 40 years), and years from diagnosis (≤ 2 vs > 2 to < 5 vs ≥ 5). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral or transdermal HRT comprising estrogen with or without progesterone for at least 2 years.
* Arm II: Patients are offered advice on nonhormonal HRT alternatives. Menopausal symptoms are assessed at baseline, at 3, 6, and 12 months, every 6 months for 4 years, and then annually thereafter. Quality of life is assessed at baseline, at 3, 6, and 12 months, every 6 months for 1 year, and then annually thereafter.

Patients are followed every 6 months for 3 years and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 2,800-3,000 patients (1,400-1,500 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Prior diagnosis of stage I or II breast cancer

  * No clinical evidence of recurrence
* Meets criteria for 1 of the following:

  * Amenorrheic for at least the past 6 months

    * Radiotherapy- or chemically-induced ovarian suppression allowed
  * Prior surgical bilateral oophorectomy
* Experiencing vasomotor symptoms (i.e., hot flashes or night sweats) with or without vaginal dryness
* No undiagnosed postmenopausal bleeding
* No ductal carcinoma in situ or lobular carcinoma in situ alone
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Postmenopausal

Sex

* Female

Menopausal status

* Postmenopausal

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* No severe, active liver disease with abnormal liver function tests
* No acute, intermittent porphyria
* Fibrinolysis and coagulation normal

Renal

* Not specified

Cardiovascular

* No prior deep vein thrombosis

  * Thrombophlebitis or superficial phlebitis alone allowed
* No prior retinal vein thrombosis

Pulmonary

* No prior pulmonary embolism

Other

* Not pregnant
* No prior alcohol, drug, or chemical abuse
* No other prior or concurrent malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* More than 3 months since prior oral or transdermal hormone replacement therapy (HRT)
* More than 5 years since prior HRT implant
* No other concurrent HRT
* No concurrent gonadotropin-releasing hormone agonists (e.g., goserelin) if less than 2 years of planned treatment remains
* No other concurrent low-dose progestins
* No concurrent tibolone
* No concurrent phytoestrogens (e.g., black cohosh, red clover, or soy)

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics

Other

* No concurrent Hypericum perforatum (St. John's wort)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: Jenni Parmar, RN — Institute of Cancer Research, United Kingdom
Locations (1):
- Institute of Cancer Research - UK, Sutton, England, United Kingdom